CLINICAL TRIAL: NCT02410265
Title: Using Technology to Address Anxiety and Stress in Indian University Students
Brief Title: Online, Guided Interventions to Reduce Generalized Anxiety Disorder Among Indian University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Craig Barr Taylor, Professor Emeritus, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31629
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Anxiety Disorders
Keywords: guided self-help; student mental health; task shifting; prevention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lantern: Guided self-help program (Experimental): Subject assigned to the Lantern intervention will receive 3-month access to a web-based, CBT-based guided self-help intervention for GAD. In the program, they receive psycho-education about GAD and the management of symptoms of GAD along with access to an "e-coach" who can monitor their progress in the program and provide feedback and encouragement via messaging and one voice call.
  Interventions: Behavioral: Lantern: Guided self-help program
- Mental Health Online: Self-help program (Experimental): Subject assigned to the Mental Health Online (MHO) intervention will receive 3-month access to a web-based, CBT-based self-help intervention for GAD. In the program, they receive psycho-education about GAD and the management of symptoms of GAD.
  Interventions: Behavioral: Mental Health Online: Self-help program
- Delayed Program (No Intervention): Subject assigned to this arm will receive one of the online programs in 9 months.

INTERVENTIONS:
Behavioral: Lantern: Guided self-help program — Subject assigned to the Lantern intervention will receive 3-month access to a web-based, CBT-based guided self-help intervention for GAD. In the program, they receive psycho-education about GAD and the management of symptoms of GAD along with access to an "e-coach" who can monitor their progress in the program and provide feedback and encouragement via messaging and one voice call.
  Arms: Lantern: Guided self-help program
Behavioral: Mental Health Online: Self-help program — Subject assigned to the Mental Health Online (MHO) intervention will receive 3-month access to a web-based, CBT-based self-help intervention for GAD. In the program, they receive psycho-education about GAD and the management of symptoms of GAD.
  Arms: Mental Health Online: Self-help program

SUMMARY:
This controlled, three-arm, randomized (1:1:1), multi-site trial will evaluate the efficacy, feasibility and acceptability of cognitive-behavioral therapy (CBT)-based online guided and unguided self-help intervention to reduce Generalized Anxiety Disorder (GAD) in Indian university students. The investigators aim to assess if these novel electronic health (eHealth) interventions can be integrated into Indian university systems to increase access to efficacious, less stigmatized, and cost-effective mental healthcare.

DETAILED DESCRIPTION:
Students from three Indian colleges will be invited to complete an online, self-report survey. Based on their answers, they are categorized into clinical, subclinical, and asymptomatic for Generalized Anxiety Disorder (GAD). Those who meet the diagnostic criteria for GAD as detailed in the Diagnostic and Statistical Manual of Mental Disorders (DSM), 4th Edition are classified as clinical. Those who score a 5.7 or above using dimensional scoring of the GAD-Q-IV but are not "clinical" are classified as subclinical. All others are asymptomatic. After ruling out those with a clinical PTSD diagnosis (scoring 38 or above on the PCL5) and those currently receiving mental healthcare treatment, those who are clinical and subclinical are offered the opportunity to use one of the online programs. Those who accept are randomized between a guided self-help program, a self-help program, and a waitlist control group. Each student who enrolls will be reassessed at post-intervention (3 months) and followup (6 months later, or 9 months after completing baseline). Additionally, those who are classified as asymptomatic are invited to complete additional followup surveys at 3 and 9 months to provide data on anxiety symptom change over time.

ELIGIBILITY:
Inclusion Criteria:

* Current student of one of the 3 college sites
* Subjects must have a clinical or subclinical diagnosis of Generalized Anxiety Disorder (GAD); clinical diagnosis is met by self-reporting DSM-IV criteria for GAD; subclinical diagnosis is met by scoring a 5.7 or above using diagnostic scoring of the GAD-Q-IV

Exclusion Criteria:

* Unable to give informed consent.
* Is currently receiving mental health treatment.
* Has clinical PTSD (a score of 38 or above on the PCL5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in GAD symptoms measured by the 4th edition of the Generalized Anxiety Disorder Questionnaire (GAD-Q-IV) | Baseline to 3-month post-intervention
  Compare GAD symptoms using the 4th edition of the Generalized Anxiety Disorder Questionnaire (GAD-Q-IV) between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.

SECONDARY OUTCOMES:
Sustained change in GAD symptoms measured by the 4th edition of the Generalized Anxiety Disorder Questionnaire (GAD-Q-IV) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare GAD symptoms using the 4th edition of the Generalized Anxiety Disorder Questionnaire (GAD-Q-IV) between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in panic disorder symptoms measured by The Panic Disorder Self-Report (PDSR) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare panic disorder symptoms using the The Panic Disorder Self-Report (PDSR) between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in social phobia symptoms measured by the Social Phobia Diagnostic Questionnaire (SPDQ) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare social anxiety disorder symptoms using the Social Phobia Diagnostic Questionnaire (SPDQ) between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in post-traumatic stress disorder symptoms measured by the Post Traumatic Stress Disorder Checklist for DSM-5 (PCL5) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare post traumatic stress disorder (PTSD) symptoms using the Post Traumatic Stress Disorder Checklist for DSM-5 between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in obsessive compulsive disorder (OCD) symptoms measured by the LEVEL 2-Repetitive Thoughts and Behaviors-Adult (adapted from the Florida Obsessive-Compulsive Inventory [FOCI] Severity Scale [Part B]) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare OCD symptoms using the the LEVEL 2-Repetitive Thoughts and Behaviors-Adult (adapted from the Florida Obsessive-Compulsive Inventory [FOCI] Severity Scale [Part B]) measure between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in specific phobia symptoms measured by questions of distress severity for specific fears | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare specific phobia symptoms using questions of distress severity for specific fears (dogs, snakes, spiders/bugs/insects, heights, flying, small enclosed spaces, driving, traveling in cars/trains/buses, bridges, tunnels, water, blood, other) between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in depression symptoms measured by the Depression Anxiety Stress Scales (DASS) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare depression symptoms using the Depression Anxiety Stress Scales (DASS) between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in worry symptoms measured by the Penn State Worry Questionnaire (PSWQ) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare worry symptoms using the Penn State Worry Questionnaire (PSWQ) between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in insomnia symptoms measured by the Insomnia Severity Index (ISI) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare insomnia symptoms using the Insomnia Severity Index between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in subject self-efficacy measured by the General Self-efficacy Scale | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare subject self-efficacy using the General Self-efficacy Scale between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in emotional distress from anxiety measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress from Anxiety measure | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare subject emotional distress from anxiety using the Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress from Anxiety measure between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in self-report difficulties with emotions, concentration, and relationships measured by the Strengths and Difficulties Questionnaire (SDQ) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare subject perception of difficulties with emotions, concentration, and relationships using the Strengths and Difficulties Questionnaire between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Change in relationship satisfaction measured by the PROMIS Satisfaction with Social Roles and Activities measure | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare subject satisfaction with social roles using the PROMIS Satisfaction with Social Roles and Activities measure between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.
Factors associated with poor program engagement and/or discontinuation measured by analysis of self-report assessments of motivation, belief in program efficacy, satisfaction, etc. as well as analysis of demographics, comorbid mental illness, etc. | Baseline to 3-month post-intervention
  Determine factors associated with poor program engagement and/or discontinuation in study participants in the guided and self-help intervention arms. Factors associated with poor program engagement and/or discontinuation will include demographics, belief in program efficacy, motivation, comorbid mental illness, socioeconomic status, and English language competence.
Change in non-specific distress measured by the Kessler Distress Measure (K10) | Baseline to 3-month post-intervention, and 6-month follow-up
  Compare subject perception of non-specific distress using the Kessler Distress measure (K10) between subjects randomized to guided self-help online programs versus self-help online programs versus waitlist control, when used for the treatment of anxiety among Indian university students with clinical and subclinical GAD.

REFERENCES:
- [Derived] Newman MG, Kanuri N, Rackoff GN, Jacobson NC, Bell MJ, Taylor CB. A randomized controlled feasibility trial of internet-delivered guided self-help for generalized anxiety disorder (GAD) among university students in India. Psychotherapy (Chic). 2021 Dec;58(4):591-601. doi: 10.1037/pst0000383. PMID 34881930
- [Derived] Kanuri N, Newman MG, Ruzek JI, Kuhn E, Manjula M, Jones M, Thomas N, Abbott JA, Sharma S, Taylor CB. The Feasibility, Acceptability, and Efficacy of Delivering Internet-Based Self-Help and Guided Self-Help Interventions for Generalized Anxiety Disorder to Indian University Students: Design of a Randomized Controlled Trial. JMIR Res Protoc. 2015 Dec 11;4(4):e136. doi: 10.2196/resprot.4783. PMID 26679295